CLINICAL TRIAL: NCT00218309
Title: Biobehavioral Studies of Opioid Drug Seeking Behavior: Study 1
Brief Title: Effects of Pre-Session Supplemental Hydromorphone on Drug Seeking Behavior in Opioid Dependent Individuals
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Wayne State University (Other)
Other Study IDs: NIDA-15462-1; R01-15462-1
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2006-05

CONDITIONS: Heroin Dependence; Opioid-Related Disorders
Keywords: opiate dependence
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders | interventions — Hydromorphone

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Hydromorphone

SUMMARY:
The purpose of this study is to determine whether the opportunity to take free supplemental hydromorphone (HYD) influences drug seeking behavior in heroin dependent individuals.

DETAILED DESCRIPTION:
Drug dependence is a condition in which drug seeking holds a higher priority than behaviors controlled by other reinforcers. Learning to understand, predict, and control this maladaptive choice behavior may lead to improved prevention and treatment strategies. HYD is a drug currently used as a cough suppressant and to relieve pain. The purpose of this study is to determine the extent to which opioid drug seeking behavior in heroin dependent individuals can be reduced by environmental factors, including supplemental opioid drug availability, drug price, and non-drug alternative reinforcers. Specifically, this study will determine whether pre-session opportunity to take "free" supplemental HYD influences HYD seeking by using a choice progressive ratio schedule as well as by varying the dose of HYD.

Participants in this observational study will undergo multiple test sessions in which they will select between acquiring drug or money. Because participants may choose money on all 12 trials of test sessions as a way to avoid receiving an injection, a placebo injection will be given when money is chosen. Prior to each test session, participants will receive a sample of the drug dose. During each test session, participants will have 12 opportunities to select either drug (administered as HYD) or money. Prior to each individual choice trial, participants will receive supplemental HYD. Participants will use a computer to earn choices. Respiration rate, oxygen saturation, heart rate, and blood pressure will be monitored throughout choice trials. Pupil diameter will be measured with a digital camera. Participants will complete self-report questionnaires at different times during the study. Participants will be maintained on buprenorphine throughout the study, with a fixed 3-week detoxification after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Current opiate dependence, verified by the structured clinical interview for DSM-IV (SCID) and Addiction Severity Index (ASI)
* Positive urine test for opiates
* Agreement to use adequate contraception for the duration of the study
* Able to read and write English

Exclusion Criteria:

* DSM-IV diagnosis of a psychiatric illness
* History of or current neurological disease, including structural brain abnormalities, seizures, infection, peripheral neuropathy, and head trauma
* History of cardiovascular disease, myocardial infarction, chest pain, edema, systolic blood pressure greater than 160 mm Hg or less than 95 mm Hg, or diastolic blood pressure greater than 95 mm Hg
* Pulmonary disease, including obstructive pulmonary disease, cor pulmonale, tuberculosis, and asthma
* Systemic diseases, such as endocrinopathies, liver or kidney failure, myxedema, hypothyroidism, Addison's disease, or autoimmune disease
* Current alcohol or sedative drug dependence
* Pregnant or breastfeeding
* Currently receiving treatment for opioid dependence
* Known phobia of injections

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16
Dates: Start 2003-09; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Derived] Woodcock EA, Lundahl LH, Burmeister M, Greenwald MK. Functional mu opioid receptor polymorphism (OPRM1 A(118) G) associated with heroin use outcomes in Caucasian males: A pilot study. Am J Addict. 2015 Jun;24(4):329-35. doi: 10.1111/ajad.12187. Epub 2015 Apr 24. PMID 25911999
- [Derived] Stoltman JJ, Woodcock EA, Lister JJ, Greenwald MK, Lundahl LH. Exploration of the telescoping effect among not-in-treatment, intensive heroin-using research volunteers. Drug Alcohol Depend. 2015 Mar 1;148:217-20. doi: 10.1016/j.drugalcdep.2015.01.010. Epub 2015 Jan 19. PMID 25630964
- [Derived] Greenwald MK, Steinmiller CL, Sliwerska E, Lundahl L, Burmeister M. BDNF Val(66)Met genotype is associated with drug-seeking phenotypes in heroin-dependent individuals: a pilot study. Addict Biol. 2013 Sep;18(5):836-45. doi: 10.1111/j.1369-1600.2011.00431.x. Epub 2012 Feb 16. PMID 22339949